CLINICAL TRIAL: NCT03180463
Title: The Study of Early Stage Osteonecrosis of Femoral Head With Human Umbilical Cord Mesenchymal Stem Cells (hUC-MSC)
Brief Title: The Study of Early Stage Osteonecrosis of Femoral Head With Human Umbilical Cord Mesenchymal Stem Cells (19#iSCLife®-ONFH)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Others
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-IMIMH-05
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Osteonecrosis of Femoral Head
Keywords: Osteonecrosis of Femoral Head; umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Core decompression surgery; Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#).
  Interventions: Drug: Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#); Procedure: core decompression
- Group 2 (Placebo Comparator): Core decompression surgery.
  Interventions: Procedure: core decompression

INTERVENTIONS:
Drug: Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#) — Allogeneic umbilical cord mesenchymal stem cells (SCLnow 19#) will be injected through surgery tunnel, 2*10^7 cells,
  Arms: Group 1
Procedure: core decompression — The surgery will drill into the femoral neck (hip bone) and through the necrotic area of the bone that died from the lack of blood flow, take out partial osseous tissue.

SUMMARY:
The purposes of the study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cells (hUC-MSC) in treating osteonecrosis of femoral head patients.

DETAILED DESCRIPTION:
This is a randomized,double-blind, paralleled study. Patients will be divided into two groups of experiment and control. All of them will receive core decompression of the femoral head, while experimental group patient will transplant hUC-MSC in addition. Follow-up visit will occur on 1 month, 3 months, and 6 months after operation, and Harris Hip score was applied to evaluate the symptoms change.

ELIGIBILITY:
Inclusion Criteria:

* Ficat classification is I, IIa, or IIb period
* no obvious improvement or ingravescence by conservative treatment
* patients or their statutory receive human umbilical cord mesenchymal stem cell of their own will, and signed informed consent form

Exclusion Criteria:

* Ficat classification is third or fourth period
* acute, chronic infection patients
* combined with heart, lung, kidney disease, and cannot tolerate operation
* ankylosing spondylitis patient
* acetabular dysplasia patient
* with tumor
* clinical data deficient
* HIV positive
* pregnancy or breast feeding women
* under other therapy that possibly influence MSC security or efficacy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI imageological examination | 6 months
  MRI imageological examination to evaluate the efficient of mesenchymal stem cells.

SECONDARY OUTCOMES:
Harris Hip Score | 6 months
  Evaluate curative effects by the change of Harris hip score.

CONTACTS AND LOCATIONS:
Overall Officials: Bahushan, Study Director — Inner Mongolia International Mongolian Hospital; Lei Guo, Dr., Study Chair — China-Japan Union Hospital, Jilin University
Locations (1):
- Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No